CLINICAL TRIAL: NCT05650489
Title: Autistic Features in Relation to Motor Function and Quality of Life in Children With an Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Other Study IDs: autism spectrum disorder
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Motor function; quality of life; autistic features
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment — correlation between Autistic features, motor function and quality of life

SUMMARY:
Although motor limitations are not currently considered a as clinical manifestation of autism spectrum disorder, should not be ignored due to their high incidence and considerable influence on life quality functional activity

ELIGIBILITY:
Inclusion Criteria:

* Both sex,
* age ranges from 3 to 5 years,
* mild to moderate autistic features according to childhood autism rating scale ,
* were able to sit alone independently

Exclusion Criteria:

* Significant visual or auditory defects,
* history of cerebral palsy or psychiatric disorder (e.g attention deficit hyperactivity disorder)

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sample size calculation was performed using G power on the correlation between childhood autism rating scale and Quality of life for Spearman's rank correlation coefficient (rs) because it was the main outcome variable in the present study. a pilot study was performed on 5 patients and showed the correlation value was (r= 0.447226 and p<0.001; and a large effect size (f= 0.447226). On the basis of the results of the pilot study (a minimum sample size of 34 patients was calculated. A sample size was increased to 34 patients, but the number will be increased to 40 to show appropriate results) a minimum sample size of 34 patients was calculated. A sample size was increased to 34 patients, but it was increased to 40 to show appropriate results.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Autism Index | baseline assessment
  Gilliam autism rating scale:
  Items on the developmental subscale address behaviors and milestones in the first 36 months of life. Items on the first three behavioral subscales are rated on a four point like scale ranging from Never Observed (0) to Frequently Observed (3). After completing it, the examiner calculated the total raw scores then converted into scaled scores and percentile ranks according to the examiner's manual. Higher scaled scores on a subscale represent severe autistic behavior. Finally, the total scaled scores were calculated to measure the autism index according to the examiner's manual. The higher the autism index, the higher the probability the individual has autism and the more severe the autistic behavior
Motor Development | baseline assessment
  The Peabody Developmental Motor Scales-Second Edition:
  The gross motor function domain will be assessed in the current study. The gross motor function domains contain four subtests. Reflexes, Stationary ,Locomotion and Object Manipulation .
  Grading and Scoring of the PDMS-2 The therapist will ask the child to do a specific item and observes how the child is doing the task. Items are scored as 2, 1 or 0.
  0 = child cannot or will not attempt an item or the attempt does not indicate that the specific skill is emerging
  * child's performance shows a clear resemblance to item mastery criteria but does not fully meet the criteria or there are signs of an emerging skill
  * child performs item according to the criteria specified for mastering the skill
Pediatric Quality of life Inventory Scale | baseline assessment
  Pediatric Quality of life Inventory Scale:
  The Arabic version will be used to assess quality of life. It contains questions about child's physical, emotional, social, and school functioning in the past 7 days. Parents/ child self-administered the quality of life after introductory instructions from the administrator. On the quality of life Generic Core Scales, for ease of interpretability, items are 22 reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better Health-Related quality of Life. To reverse score, transform the 0-4 scale items to 0-100 as follows: 0-100, 1=75, 2= 50, 3= 25 and 4= 0. Finally, the Scale Score for each dimension and Total Scale Score were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Eman s Albadry, B.S.C, Principal Investigator — Cairo university, faculty of physical therapy; Amr A OTHMAN, Principal Investigator — Sohag University; MAI E ABBASS, Study Chair — Cairo university, faculty of physical therapy
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt